CLINICAL TRIAL: NCT03029169
Title: Prospective Randomized Study of Efficacy and Safety of 1c Class Antiarrhythmic Agent (Propafenone) in Septic Shock
Brief Title: Propafenone Versus Amiodarone in Septic Shock
Acronym: PRASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Martin Balik, A/Prof, MD, PhD, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1691/16 S-IV
Record Dates: First submitted 2016-12-07; First posted 2017-01-24 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Supraventricular Arrhythmia; Septic Shock
Keywords: Supraventricular Arrhythmia; Septic shock; Propafenone; Amiodarone; Intensive Care
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Provided by a dedicated study nurse
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propafenone i.v. (Active Comparator): Patients in septic shock with a new onset supraventricular arrhythmia are randomized either to arm treated with propafenone or with amiodarone. Both arms will have standard treatment, there are no limits to indicated electric cardioversion as part of treatment.
  Intervention: Bolus of 35-70 mg intravenous propafenone followed by continuous infusion of 400-840 mg/24h.
  Interventions: Drug: Propafenone i.v.
- Amiodarone i.v. (Active Comparator): Patients in septic shock with a new onset supraventricular arrhythmia are randomized either to arm treated with propafenone or with amiodarone. Both arms will have standard treatment, there are no limits to indicated electric cardioversion as part of treatment.
  Intervention: Bolus of 150-300 mg of intravenous amiodarone followed by continuous infusion of 600-1800 mg/24h.
  Interventions: Drug: Amiodarone i.v.

INTERVENTIONS:
Drug: Propafenone i.v. — Treatment
  Other Names: Antiarrhythmic therapy
  Arms: Propafenone i.v.
Drug: Amiodarone i.v. — Treatment
  Other Names: Antiarrhythmic therapy
  Arms: Amiodarone i.v.

SUMMARY:
Arrhythmias accompany septic shock in increased rates than in other ICU cohorts and their presence and management are related to patient´s prognosis. 1c class antiarrhythmics are seldom administered in intensive care due to a dose dependent toxicity published in case reports and unfavourable outcome reported in a few prospective trials done on cardiology patients. The papers on 1c class antiarrhythmics do not take into consideration a complex haemodynamic assessment using echocardiography. The authors have recently presented a retrospective study on SV arrhythmias in septic shock patients demonstrating favourable effect and safety of propafenone which showed higher antiarrhythmic efficacy than amiodarone.

DETAILED DESCRIPTION:
Primary aim is to verify the conclusions of the retrospective study, i.e. efficacy and safety of propafenone, in a prospective blinded randomized trial performed in two large intensive care units. Secondary aims are to monitor the electromechanics of left atrium in patients with SV arrhythmias in septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock with a new onset SV arrhythmia
* LV systolic function normal to moderately reduced according to echocardiography.

Exclusion Criteria:

* Severe LV systolic dysfunction
* More than 1st degree AV block
* High dose vasopressor therapy with continuous noradrenaline > 1.0 ug/kg.min
* Known intolerance to amiodarone or propafenone
* Absence of septic shock
* Chronic AF
* Dependence on pacemaker
* Status after MAZE procedure

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of propafenone | 1 year
  cardioversion rate
ICU mortality of septic shock patients on propafenone for a SV arrhythmia | 1 year
  ICU mortality
28-day mortality of septic shock patients on propafenone for a SV arrhythmia | 2 years
  28-day mortality
12-month mortality of septic shock patients on propafenone for a SV arrhythmia | 2 years
  12-month mortality

SECONDARY OUTCOMES:
Electromechanics of left atrium | 1 year
  left atrial emptying
Electromechanics of LA | 1 year
  isovolumic and ejection times

CONTACTS AND LOCATIONS:
Overall Officials: Martin Balik, A/Prof, Principal Investigator — Dept of Anaesthesia and Intensive Care
Locations (2):
- Czechia (2):
  - Dept. Anaesthesia and Intensive Care, 3rd Medical Faculty, Charles University, Prague
  - Dept of Anaesthesia and Intensive Care, General University Hospital, 1st Medical Faculty, Charles University, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balik M, Waldauf P, Maly M, Brozek T, Rulisek J, Porizka M, Sachl R, Otahal M, Brestovansky P, Svobodova E, Flaksa M, Stach Z, Horejsek J, Volny L, Jurisinova I, Novotny A, Trachta P, Kunstyr J, Kopecky P, Tencer T, Pazout J, Krajcova A, Duska F. Echocardiography predictors of sustained sinus rhythm after cardioversion of supraventricular arrhythmia in patients with septic shock. J Crit Care. 2024 Oct;83:154832. doi: 10.1016/j.jcrc.2024.154832. Epub 2024 May 17. PMID 38759581
- [Derived] Waldauf P, Porizka M, Horejsek J, Otahal M, Svobodova E, Jurisinova I, Maly M, Brozek T, Rulisek J, Trachta P, Tencer T, Krajcova A, Duska F, Balik M. The outcomes of patients with septic shock treated with propafenone compared to amiodarone for supraventricular arrhythmias are related to end-systolic left atrial volume. Eur Heart J Acute Cardiovasc Care. 2024 May 28;13(5):414-422. doi: 10.1093/ehjacc/zuae023. PMID 38372622
- [Derived] Balik M, Waldauf P, Maly M, Matousek V, Brozek T, Rulisek J, Porizka M, Sachl R, Otahal M, Brestovansky P, Svobodova E, Flaksa M, Stach Z, Pazout J, Duska F, Smid O, Stritesky M. Efficacy and safety of 1C class antiarrhythmic agent (propafenone) for supraventricular arrhythmias in septic shock compared to amiodarone: protocol of a prospective randomised double-blind study. BMJ Open. 2019 Sep 3;9(9):e031678. doi: 10.1136/bmjopen-2019-031678. PMID 31481571